CLINICAL TRIAL: NCT01367808
Title: Effects of Posaconazole and Voriconazole on the Pharmacokinetics and Pharmacodynamics of Sublingual Buprenorphine: A Three-phase Cross-over Study in Healthy Subjects
Brief Title: Effects of Posaconazole and Voriconazole on the Pharmacokinetics and Pharmacodynamics of Sublingual Buprenorphine
Acronym: PosaBupre
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Professor Klaus T Olkkola, Department of Anaesthesiology & Intensive Care
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 55/180/2010
Record Dates: First submitted 2011-05-30; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2010-12

CONDITIONS: Pharmacokinetics and Pharmacodynamics of Sublingual Buprenorphine
Keywords: Buprenorphine; Vorikonazole; Posakonazole; Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vorikonazole (Active Comparator)
  Interventions: Drug: vorikonazole
- Posakonazole (Active Comparator)
  Interventions: Drug: posakonazole

INTERVENTIONS:
Drug: Placebo — The subjects will be given placebo twice a day for 5 days prior to the study
  Arms: Placebo
Drug: vorikonazole — The subject will be given vorikonazole twice a day for 5 days prior to the study. The dose will be 400 mg twice a day on day one ans 200 mg twice a day on days 2-5.
  Arms: Vorikonazole
Drug: posakonazole — The subjects will be given posaconazole 400 mg twice a day for 5 days prior to the study.
  Arms: Posakonazole

SUMMARY:
Variability in drug response can be due to either pharmacokinetic or pharmacodynamic factors. The reasons why people differ in pharmacokinetics or pharmacodynamics are manifold and include, e.g., genetic factors, diseases, age and concomitantly administered drugs. Oxidation reactions are dominant in the metabolism of drugs and cytochrome P-450 enzymes (CYP) have been recognized as chief contributors. We have previously shown that drug interactions mediated by the inhibition of CYP enzymes may be of major clinical significance.

This study is aimed to examine the possible interactions of low-dose sublingual buprenorphine with posaconazole and voriconazole.

The study will be conducted using a randomized, balanced cross-over design in three phases.

Twelve male or female adult non-smoking subjects aged 18-40 years with body weights within ±15% of the ideal weight for height will be recruited for the study. The subjects will be submitted to physical examination, determination of previous or present chronic diseases, and comprehensive laboratory testing to ascertain that they are in good health. The subjects will fill in a modified Finnish version of the Abuse Questions to assess their vulnerability for opioid abuse. Laboratory screening will include CBC (including hemoglobin, hematocrit, differential WBC, platelet count), SGOT, SGPT, alkaline phosphatase, BUN and creatinine, and for women a pregnancy test. Urine will be screened for glucose, proteins and drugs with addiction potential. Blood pressure in sitting position must be within normal limits. Base line ECG must be normal.

The subjects will be given in a randomized, cross-over, balanced manner at intervals of four weeks either placebo, vorikonazole or posakonazole. On day 5, the challenge dose of 0.4 or 0.6 mg of sublingual buprenorphine (Temgesic, Schering-Plough) will be administered at 11.00, i.e. 1 h after the last dose of placebo, voriconazole or posaconazole. The dose is 0.6 mg after placebo and 0.4 mg after posaconazole and voriconazole. If necessary, naloxone (Naloxone B. Braun, Braun) will be given in sufficient doses to counteract the severe adverse effects of buprenorphine. For nausea and vomiting, intravenous tropisetron will used, if needed.

On day 4, a forearm vein will be cannulated with a plastic cannula for blood sampling. Timed venous blood samples will be drawn before the administration of buprenorphine and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 18-20 hours after administration. Another venous cannula will be inserted to the opposite forearm for the intravenous administration of naloxone. Urine will be collected for 18-20 hours.

The psychomotor effects of buprenorphine will be assessed with visual analog scales (Bond and Lader 1974) and digit symbol substitution test (Stone 1984) at 1-2 hour intervals up to 12 hours after buprenorphine administration. Visual analogue scales will be used for the following items: alert / drowsy, good / poor performance, no / strong drug effect, unpleasant /pleasant feeling, no / extreme nausea. For each pharmacodynamic variable, the area under the response-time curve will be determined by trapezoidal rule for 12 hours.

The analgesic effect of buprenorphine will be evaluated using the cold pressor test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-40
* Body weight within ±15% of the ideal weight for height

Exclusion Criteria:

* A previous history of intolerance to the study drugs or to related compounds and additives
* Concomitant drug therapy of any kind for at least 14 days prior to the study
* Existing or recent significant disease
* History of hematological, endocrine, metabolic or gastrointestinal disease, including gut motility disorders
* History of asthma or any kind of drug allergy
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements
* A positive test result for urine toxicology
* A "yes" answer to any one of the Abuse Questions
* Pregnancy or nursing
* Donation of blood for 4 weeks prior and during the study
* Special diet or life style conditions which would compromise the conditions of the study or interpretation of the results
* Participation in any other studies involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study
* Smoking for one month before the start of the study and during the whole study period
* Any history of coagulation abnormality, also in first degree relatives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Concentration of buprenorphine and its metabolites in plasma and urine | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 20 hours after administration of buprenorphine

SECONDARY OUTCOMES:
Pharmacodynamic effects | 1, 2,3, 4, 5, 6, 8, 10, 12, hours after administration of buprenorphine
  The psychomotor effects on buprenorphine will be assessed with the measurement of pupil size, Maddox wing test and digit symbol substitution test
Analgesia | 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after the administration of buprenorphine
  The analgesic effect of buprenorphine will be evaluated using the cold pressor test. Briefly, the subject's hand is immersed into ice-cold water of + 4° C up to the wrist. The subject is told to keep his or her hand in the water and to report when the cold sensation becomes painful. Cold pain threshold is defined as the latency from the immersion of the hand to the subject's first report of pain. Cold pain intensity is assessed at 30 s intervals following immersion of the hand in cold water for up to 60s . A verbal numerical rating scale of 0-100 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus T Olkkola, professor, Principal Investigator — Turku University Hospital
Locations (1):
- Department of Anaesthesiology & Intensive Care, Turku, Finland